CLINICAL TRIAL: NCT00001688
Title: A Pilot Study of the Immunologic Reconstitution in HIV-1 Infected Children Receiving Highly Active Antiretroviral Therapy With Combination Ritonavir, Nevirapine and Stavudine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980041; 98-C-0041
Record Dates: First submitted 1999-11-03; First posted 2002-05-22 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-11

CONDITIONS: HIV Infection
Keywords: CD4 Cells; Cytokines; Anti-Retroviral Activity; V Beta Repertoire; CD-4-Naive T Cells; CD-4-Memory T Cells
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nevirapine; Stavudine

INTERVENTIONS:
Drug: Ritonavir
Drug: Nevirapine
Drug: Stavudine

SUMMARY:
This is a pilot study to evaluate the ability of highly active antiretroviral therapy administered to children with HIV-1 infection to effect immunoreconstitution in children with HIV-1 infection. In addition, this study will determine the safety of combination therapy with ritonavir, nevirapine and stavudine (d4T) as well as the anti-HIV activity of combination therapy with ritonavir, nevirapine and stavudine. A total of 25 HIV-1 infected children will be studied, including both moderately and severely immunocompromised individuals. The children will be treated with ritonavir, nevirapine and stavudine or with predefined drug substitutions in the case of intolerance. Immunoreconstitution, defined as the repopulation of naive T cells, will be studied by determining the presence and extent of production of new naive (thymic derived) CD4+ T cells and their T cell receptor repertoire. Drug pharmacokinetic profiles in this regimen will be examined.

DETAILED DESCRIPTION:
This is a pilot study to evaluate the ability of highly active antiretroviral therapy administered to children with HIV-1 infection to effect immunoreconstitution in children with HIV-1 infection. In addition, this study will determine the safety of combination therapy with ritonavir, nevirapine and stavudine (d4T) as well as the anti-HIV activity of combination therapy with ritonavir, nevirapine and stavudine. A total of 25 HIV-1 infected children will be studied, including both moderately and severely immunocompromised individuals. The children will be treated with ritonavir, nevirapine and stavudine or with predefined drug substitutions in the case of intolerance. Immunoreconstitution, defined as the repopulation of naive T cells, will be studied by determining the presence and extent of production of new naive (thymic derived) CD4+ T cells and their T cell receptor repertoire. Drug pharmacokinetic profiles in this regimen will be examined.

ELIGIBILITY:
Children between ages of 4 years and 18 years.

Diagnosis of HIV-1 infection as defined by the Centers for Disease Control (CDC) Definition.

Availability of a parent or guardian to provide Informed Consent.

Child is not critically ill or clinically unstable.

No CDC categories N1 and A1 (1994 revised classification for HIV infection in children less than 13 years of age) and the CDC 1993 revised HIV classification and expanded AIDS surveillance definition for adolescents and adults.

Non-presence of an active opportunistic infection requiring acute intervention at the time of entry (e.g. CMV, aspergillosis, cryptococcosis, Candida, etc.). Patients receiving treatment for an infection that requires prolonged treatment must have been stable on therapy for at least 30 days prior to study entry.

No administration of chemotherapeutic agents, investigational agents or use of immunomodulating agents such as IVIG, corticosteroids, interferons, pentoxifylline, G-CSF/GM-CSF, erythropoeitin, growth hormone and other growth factors within one month of enrollment.

None of the following laboratory abnormalities within 2 weeks of study entry:

Total WBC count less than 1500/mm(3) or an absolute neutrophil count less than 750/mm(3);

Hemoglobin less than 8.0 g/dl;

Platelet count less than 75,000/mm(3);

Creatinine greater than 2.0 x normal;

Creatinine clearance less than or equal to 50 mL/min/m(2);

Total bilirubin greater than 2 x normal;

SGOT/SGPT greater than 5 x normal;

Serum amylase pancreatic isoenzyme greater than 90 U/L (2 x upper limit of normal for adult). Serum amylase pancreatic isoenzyme should be obtained only if total serum amylase is greater than 180 U/L.

No history of clinical pancreatitis and/or elevation in serum amylase pancreatic isoenzyme of greater than 180 U/L.

No history of peripheral neuropathy of Grade II or greater severity.

No previous treatment with ritonavir, indinavir, nelfinavir, nevirapine or stavudine. Patients may have received treatment with ritonavir, indinavir, nelfinavir for less than 4 weeks.

Ability to swallow tablets.

No child for whom the volume of research blood required for study evaluation exceeds the maximum volume of research blood allowable (3 ml/kg in a single blood withdrawal and 7 ml/kg in a 6-week period). This would be applicable to a child less than 16.5 kg.

No patients who refuse or cannot have leukapheresis done.

Sexually active post-menarchal females must be willing to use a barrier method of contraception or be willing to remain sexually abstinent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1998-01; Study Completion 2001-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Yarchoan R, Mitsuya H, Broder S. Challenges in the therapy of HIV infection. Immunol Today. 1993 Jun;14(6):303-9. doi: 10.1016/0167-5699(93)90050-U. PMID 8397771
- [Background] Mackall CL, Granger L, Sheard MA, Cepeda R, Gress RE. T-cell regeneration after bone marrow transplantation: differential CD45 isoform expression on thymic-derived versus thymic-independent progeny. Blood. 1993 Oct 15;82(8):2585-94. PMID 7691265
- [Background] Mackall CL, Fleisher TA, Brown MR, Andrich MP, Chen CC, Feuerstein IM, Horowitz ME, Magrath IT, Shad AT, Steinberg SM, et al. Age, thymopoiesis, and CD4+ T-lymphocyte regeneration after intensive chemotherapy. N Engl J Med. 1995 Jan 19;332(3):143-9. doi: 10.1056/NEJM199501193320303. PMID 7800006